CLINICAL TRIAL: NCT02691403
Title: Ultrasound-guided Quadratus Lumborum Block for Postoperative Analgesia After Colostomy: A Randomized Controlled Trial
Brief Title: Quadratus Lumborum Block for Postoperative Analgesia After Colostomy Closure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Nai Liang Li, Doctor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QLCO
Record Dates: First submitted 2016-02-17; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Placebo QL block (Sham Comparator): 30 ml single shot QL block with saline 0.9%
  Interventions: Drug: normal saline
- Active QL block (Active Comparator): 30 ml single shot QL block with 0.25% levo-bupivacaine
  Interventions: Drug: levo-bupivacaine

INTERVENTIONS:
Drug: levo-bupivacaine
  Arms: Active QL block
Drug: normal saline
  Arms: Placebo QL block

SUMMARY:
Patients undergoing abdominal procedures often require multimodal postoperative pain controls. Truncal blocks such as quadratus lumborum (QL) block may be used adjunctively as a part of it. The investigators hypothesized that the ultrasound-guided QL block with transmuscular approach can provide adequate pain relief for colostomy closure as part of a multimodal pain control.

ELIGIBILITY:
Inclusion Criteria:

* A physical status between ASA I and III
* 20 - 75 years of age
* Patient has signed an informed consent
* Without contraindication of QL block

Exclusion Criteria

* American Society of Anesthesiologists (ASA) Physical Status ≥ 4
* Any contraindication to nerve blocks (including coagulopathy, abnormal anatomy, infection at the planned QL injection site, and amide-type local anesthetic allergy) pregnancy or breast-feeding
* Severe obesity (body mass index≥ 35 kg/m2)
* Patients with a history of significant neurological, psychiatric, neuromuscular, cardiovascular, pulmonary, renal or hepatic disease
* Allergy to NSAIDs
* Infection at the QL injection site
* Patients with major psychosis or drug and alcohol abuse
* Patient unable to comprehend or use the verbal rating pain scoring system or patient-controlled analgesia pump

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
cumulative morphine consumption | 1 hour